CLINICAL TRIAL: NCT02595515
Title: The Effect of Chiropractic Treatment of Infantile Colic. A Randomized, Controlled Trial
Brief Title: The Effect of Chiropractic Treatment of Infantile Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Institute of Chiropractic and Clinical Biomechanics (Other)
Collaborators: Research Unit of General Practice, Odense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: -14/1206
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chiropractic treatment (Experimental): Manipulation and/or mobilisation. Intervention: Procedure: Chiropractic treatment.
  Interventions: Other: Chiropractic treatment
- Visit without active treatment (Placebo Comparator): The child is brought in for chiropractic treatment, but no active treatment is delivered. The parents are unaware whether the treatment is delivered or not.
  Interventions: Other: Visit without active treatment

INTERVENTIONS:
Other: Chiropractic treatment — Procedure: chiropractic treatment.
  Other Names: Manipulation; mobilisation
  Arms: Chiropractic treatment
Other: Visit without active treatment — Procedure: Visit without active treatment. The child is brought in for chiropractic treatment, but no active treatment is delivered. The parents are unaware whether the treatment is delivered or not.
  Arms: Visit without active treatment

SUMMARY:
Infantile colic is condition that affects more than 10% of babies and their families. The reason, and hence proper treatment, for this condition is unknown and many causes have been suggested. One of the treatments that parents choose is chiropractic manipulation. In Denmark, almost 10,000 babies are each year treated by chiropractors, and a high proportion is due to colic. However, the effect of chiropractic treatment of infantile colic has not been properly scientifically evaluated.

The effects of chiropractic treatment on infantile colic needs to be investigated, since this is a very common disorder with no known effective treatment, but with good empirical evidence of the value of chiropractic treatment. Although it is usually considered to be a benign and self-limiting condition, some studies suggest there might be long-term effects in terms of psychomotor problems. In worst case, the infants' crying may also lead to violence and 'shaken baby syndrome'.

Null hypothesis: There is no effect of chiropractic treatment on the course of infantile colic.

This study is a controlled, clinical trial where infants fulfilling the diagnostic criteria for colic will be randomized into two groups. One group will receive treatment and the other won't. This will determine the overall effect and furthermore, subgroup analyses will be performed to identify possible subgroups of infants, who will benefit the most from the treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary: To investigate the effect of chiropractic treatment on infantile colic

Secondary: to investigate if infants with suspected musculoskeletal problems respond differently to the treatment than those without.

METHOD:

A randomized controlled single blind multicenter clinical trial

The project is to be carried out on the island of Funen, Denmark. Recruitment of babies with symptoms of infantile colic is based on contact by the parents of the babies to the project manager. Information about the existence of the study is given to health visitors, general practitioners, midwifes and to women who have given birth on the maternity ward in the University Hospital of Odense. For infants fulfilling the diagnostic criteria for colic the parents will register amount of crying using a valid instrument for at least three days before the first visit at the chiropractor Clinic (baseline registration). The babies will be randomized to chiropractic treatment or no treatment. The parents will be unaware of the child's allocation. All children have four visits during two weeks at the chiropractor. All children will be taken to the chiropractor's treatment room, while the parents stay in the reception areas. Before treatment, the chiropractors will note, whether they suspect musculoskeletal involvement or not. The parents register the amount of crying continuously during the two weeks and up to and including three days after the fourth visit. Three days after the the fourth visit, the parents are informed by the chiropractor about the child's allocation. Children in the control group will afterwards have the opportunity to have four free visits with chiropractic treatment.

The parents will be asked to give consent that the medical journal regarding pregnancy and birth is reviewed in order to obtain information on specific measures (e.g. duration of pregnancy, duration of labor, delivery presentation, vacuum extractor delivery or caesarean section). Subgroup analyses will be performed to investigate associations with symptoms of colic and suspected musculoskeletal involvement. All analyses will be adjusted for known confounders, registered by the project manager at baseline.

PERSPECTIVE FOR HEALTHCARE:

First of all, the study will evaluate the effect of chiropractic treatment of infantile colic. Secondly, it will clarify if the treatment effect differs between children with suspected musculoskeletal involvement and those without.

ELIGIBILITY:
Inclusion Criteria:

* Age: 2-14 weeks.
* Minimum crying and fussing: three hours per day, three days per week
* Satisfying weight gain

Exclusion Criteria:

* Known disease
* Symptoms than can indicate other condition than infantile colic
* Contraindications for chiropractic treatment
* Previous chiropractic treatment due to infantile colic

Ages: 2 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2015-11; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in hours of crying | Two weeks
  Change in number of crying hours per day based on parental diaries (before and after treatment) when comparing treated and not treated children

SECONDARY OUTCOMES:
Change in hours of crying for children with suspected musculo-skeletal problems | Two weeks
  Subgroup analysis for the children with suspected musculo-skeletal problems including change in number of crying hours per day based on parental diaries (before and after treatment) when comparing treated and not treated children

CONTACTS AND LOCATIONS:
Overall Officials: Lise V Holm, MD, PhD, Principal Investigator — Research Unit of General Practice, Odense, University of Southern Denmark, JB Wilsløwsvej 9A, 5000 Odense C, Denmark; Lise Hestbæk, Assoc Prof, Study Director — Nordic Institute of Chiropractic and Clinical Biomechanics. Campusvej 55, 5250 Odense M, DK, Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Holm LV, Vach W, Jarbol DE, Christensen HW, Sondergaard J, Hestbaek L. Identifying potential treatment effect modifiers of the effectiveness of chiropractic care to infants with colic through prespecified secondary analyses of a randomised controlled trial. Chiropr Man Therap. 2021 Apr 19;29(1):16. doi: 10.1186/s12998-021-00373-6. PMID 33874964
- [Derived] Holm LV, Jarbol DE, Christensen HW, Sondergaard J, Hestbaek L. The effect of chiropractic care on infantile colic: results from a single-blind randomised controlled trial. Chiropr Man Therap. 2021 Apr 19;29(1):15. doi: 10.1186/s12998-021-00371-8. PMID 33874955
- [Derived] Holm LV, Jarbol DE, Christensen HW, Sondergaard J, Hestbaek L. The effect of chiropractic treatment on infantile colic: study protocol for a single-blind randomized controlled trial. Chiropr Man Therap. 2018 Jun 7;26:17. doi: 10.1186/s12998-018-0188-9. eCollection 2018. PMID 29930798